CLINICAL TRIAL: NCT04412421
Title: Adherence to Vitamin and Mineral Supplementation After Bariatric Surgery
Brief Title: Supplementation After Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ellen Andersson, MD, PhD, Consultant Upper GI Surgeon, Region Östergötland
Other Study IDs: Vitamin study 01
Record Dates: First submitted 2020-02-07; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Bariatric Surgery; Micronutrient Deficiencies; Obesity
Keywords: Bariatric Surgery (Gastric Bypass, Gastric Sleeve); Micronutrient Deficiencies; Adherence, Medication
MeSH Terms: conditions — Obesity; Medication Adherence | interventions — Gastric Bypass; Vitamins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Gastric Bypass, Sleeve Gastrectomy — Lifelong vitamin and Mineral supplementation
  Other Names: Vitamin and Mineral supplementation

SUMMARY:
The aim of this study is to assess medication adherence to vitamin and mineral supplements after bariatric surgery and identify factors that may influence adherence. All study participants are prescribed life-long treatment with daily oral vitamin B12 and Calcium/Vitamin-D. Menstruating women are also prescribed daily oral iron supplementation. Post-operative adherence rate is retrieved from Pharmacy refill data, collected from the Swedish Prescribed Drug Register, the five first years after bariatric surgery.

DETAILED DESCRIPTION:
The aim of this study is to assess medication adherence to vitamin- and mineral supplementation after bariatric surgery, identify factors that may influence adherence, as well as study the development of micronutrient deficinencies detectable by blood sampling.

All study participants are prescribed life-long treatment with daily oral vitamin B12 and Calcium/Vitamin-D. Menstruating women are also prescribed daily oral iron supplementation.

Post-operative adherence rate is retrieved from pharmacy refill data, collected from The Swedish Prescribed Drug Register, at one, two and five years after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients subjected to bariatric surgery at Vrinnevi Hospital, Norrköping, Sweden

Exclusion Criteria:

* Unable to read and understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients subjected to bariatric surgery at Vrinnevi Hospital
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to vitamin and mineral supplementation | 5 years
  Implementation (Continuous multiple-interval measures of medication availability/gaps, CMA),
Time to initiation | 1 year
  Initiation (time to initiation)
Time to discontinuation | 5 years
  Discontinuation (Time to discontinuation)

SECONDARY OUTCOMES:
Self reported Adherence to vitamin-and mineral supplementation | 5 years
  Medication Adherence Report Scale (MARS-5) score 1-25, higher scores mean a better outcome
Hemoglobin (Hb) | 5 years
  g/L
Iron status | 5 years
  µmol/L
s-folate | 5 years
  nmol/L
p-calcium | 5 years
  mmol/L
s-albumin | 5 years
  g/L
s-cobolamin | 5 years
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Andersson, Principal Investigator — Region Östergötland
Locations (1):
- Department of Surgery, Vrinnevi Hospital, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No